CLINICAL TRIAL: NCT00284180
Title: Phase II Trial of Vinflunine Plus Trastuzumab in Human Epidermal Growth Factor Receptor 2 (HER2neu) Over-Expressing Metastatic Breast Cancer
Brief Title: Vinflunine Plus Trastuzumab in Human Epidermal Growth Factor Receptor 2 (HER2neu) Over-Expressing Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCRI BRE 89
Record Dates: First submitted 2006-01-27; First posted 2006-01-31 (Estimated); Results first posted 2013-08-09 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-07

CONDITIONS: Breast Neoplasms; Breast Cancer
Keywords: Breast Neoplasms; Breast Cancer; Vinflunine; Vinca Alkaloid; Javlor
MeSH Terms: conditions — Breast Neoplasms | interventions — vinflunine; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HER2 Negative Intervention (Experimental): Vinflunine 320 mg/m2 intravenously day 1 over 20 minutes, repeated every 21 days
  Interventions: Drug: Vinflunine
- HER2 Positive Intervention (Experimental): Vinflunine 280 mg/m2 every 21 days with trastuzumab administered with a loading dose of 8 mg/kg, followed by 6 mg/kg IV on day 1 of each subsequent cycle, repeated every 21 days. If no grade 3/4 adverse events were encountered after the first cycle of vinflunine/trastuzumab, the dose of vinflunine could be escalated to 320 mg/m2.
  Interventions: Drug: Vinflunine; Drug: Trastuzumab

INTERVENTIONS:
Drug: Vinflunine — Novel second generation vinca alkaloid
  Other Names: Javlor
Drug: Trastuzumab — Anti-HER2 monoclonal antibody
  Other Names: Herceptin
  Arms: HER2 Positive Intervention

SUMMARY:
This research study involves the anti-cancer medication trastuzumab and the investigational drug vinflunine. The purpose of this trials is to see if trastuzumab and vinflunine used in combination or vinflunine alone is effective in the treatment of metastatic breast cancer

DETAILED DESCRIPTION:
If the tumor is HER2neu positive, eligible patients will receive trastuzumab and vinflunine intravenously (IV) every 3 weeks.

If the tumor is HER2neu negative, eligible patients will receive vinflunine intravenously (IV) every 3 weeks.

Patients whose cancer does not grow or decreases in size may continue to receive treatment until cancer progression. Evaluation of cancer will be every 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed breast cancer with metastatic disease. Patients without pathologic or cytologic confirmation of metastatic disease should have unequivocal evidence of metastasis using the Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* The human epidermal growth factor receptor 2 (HER2) status of the tumor will be used to stratify patients. Tumors that are HER2 FISH+ will receive vinflunine and trastuzumab. Patients with tumors which are HER2 FISH negative or if the HER2 status is unknown/not performed will remain on study and will receive single agent vinflunine.
* Patients must have measurable disease not directly irradiated as per RECIST criteria.
* Measurable disease- is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan.
* Prior Therapy: Patients must not have received prior chemotherapy in the metastatic breast setting. Patients who have not received prior anthracyclines or taxanes should be considered for these agents. Patients may have received prior chemotherapy and/or hormonal therapy for early stage breast cancer. The chemotherapy regimen may have included an anthracycline and/or a taxane as long as it has been > 6 months since completion of the regimen. Adjuvant trastuzumab is allowed. Patients may have received prior radiation therapy in either the metastatic or early stage setting as long as <25% of the bone marrow has been treated. Prior radiation to the whole pelvis is not allowed. Radiation therapy must be completed at least 7 days prior to study registration, and all radiation related toxicities must be resolved to grade ≤ 1 before patient is eligible for study inclusion. Patients may have received any number of hormonal therapies in the neo-adjuvant, adjuvant or metastatic setting.
* Age >18 years.
* Life expectancy of > 6 months.
* Eastern Cooperative Oncology Group (ECOG) performance status <2.
* Patients must have normal organ and marrow function. Laboratory tests should be completed within 14 days prior to starting study treatment. Only for patients who will be receiving trastuzumab, a left ventricular ejection fraction (LVEF) may be determined by either echocardiography or multigated acquisition (MUGA) scan, and should be obtained within 4 weeks prior to starting study treatment.
* Fertility/reproduction. Patients must not be pregnant, expect to become pregnant or conceive a child from time of first signing study consent until at least 12 weeks after last dose of study treatment.

Exclusion Criteria

* Patients who have received prior vinca alkaloid chemotherapy are not eligible unless treatment was completed > 5 years ago.
* Patients in which the HER2 status is unknown or is FISH negative will not receive trastuzumab but are eligible for treatment with single agent vinflunine.
* Patients that have received prior chemotherapy for metastatic breast cancer.
* Patients receiving trastuzumab must have received a cumulative dose of doxorubicin less than 360mg/m2, and/or an epirubicin cumulative dose less than 720mg/m2 for study entry.
* Patients with known leptomeningeal carcinomatosis are excluded from this clinical trial
* History of grade 3 or 4 allergic reactions attributed to trastuzumab.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study
* History of other non-breast cancer malignancy except for carcinoma in situ of the cervix or non-melanoma skin cancer, or in patients with greater than a 5-year disease free interval from a prior malignancy.
* Patients who have received prior chemotherapy for early stage breast cancer with the completion of the regimen being < 6 months will not be eligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-01; Primary Completion 2008-02 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise A Yardley, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (10):
- United States (10):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Florida Cancer Specialists, Fort Myers, Florida
  - Integrated Community Oncology Network, Jacksonville, Florida
  - Watson Clinic Center for Cancer Care and Research, Lakeland, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Hematology Oncology Life Center, Alexandria, Louisiana
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Associates in Hematology Oncology, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee

REFERENCES:
- [Result] Yardley DA, McCleod M, Schreiber F, Murphy P, Patton J, Thompson DS, Shastry M, Rubin M, Melnik M, Burris HA, Hainsworth JD. A phase II trial of vinflunine as monotherapy or in combination with trastuzumab as first-line treatment of metastatic breast cancer. Cancer Invest. 2010 Nov;28(9):925-31. doi: 10.3109/07357907.2010.496755. PMID 20690806
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/20690806

RESULTS

PARTICIPANT FLOW:
Groups:
- Vinflunine: Vinflunine 320 mg/m2 intravenously day 1 over 20 minutes repeated every 21 days
- Vinflunine/Trastuzumab: Vinflunine 280 mg/m2 every 21 days with trastuzumab administered with a loading dose of 8 mg/kg, followed by 6 mg/kg IV on day 1 of each subsequent cycle, repeated every 21 days. If no grade 3/4 adverse events were encountered after the first cycle, the dose could be escalated to 320 mg/m2
Period: Overall Study
Arm/Group | Vinflunine | Vinflunine/Trastuzumab
Started | 11 | 21
Completed | 11 | 17
Not Completed | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vinflunine | Vinflunine/Trastuzumab | Total
Number analyzed (Participants) | 11 | 21 | 32
Age Continuous [Median (Full Range); unit: years] | 59 [47 to 78] | 58 [35 to 78] | 59 [35 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 21 | 32
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 21 | 32

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR), the Percentage of Patients Who Experience an Objective Benefit From Treatment
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 18 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Vinflunine/Trastuzumab: Vinflunine 280 mg/m2 every 21 days with trastuzumab administered with a loading dose of 8 mg/kg, followed by 6 mg/kg IV on day 1 of each subsequent cycle, repeated every 21 days. If no grade 3/4 adverse events were encountered after the first cycle of vinflunine/trastuzumab, the dose of vinflunine could be escalated to 320 mg/m2
Arm/Group | Vinflunine | Vinflunine/Trastuzumab
Number analyzed (Participants) | 11 | 21
percentage of participants | 9 [0.23 to 41.26] | 33 [14.59 to 56.97]

ADVERSE EVENTS:
Arm/Group | Vinflunine | Vinflunine/Trastuzumab
Serious Adverse Events (participants affected / at risk) | 5/11 | 8/21
Other Adverse Events (participants affected / at risk) | 11/11 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vinflunine (N=11) | Vinflunine/Trastuzumab (N=21)
Progressive Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dehydration (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Right femur
CNS Ischemia (Nervous system disorders) | 1 (1) | 1 (1)
Pain NOS (General disorders) | 2 (2) | 0 (0) — Pain not otherwise specified
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diabetes insipidus (Endocrine disorders) | 1 (1) | 0 (0) — Diabetes Insipidus
Thrombosis/Thrombus/Embolism (Vascular disorders) | 1 (1) | 0 (0)
Pain - abdomen (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vinflunine (N=11) | Vinflunine/Trastuzumab (N=21)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (13) | 5 (30)
Anorexia (Gastrointestinal disorders) | 4 (9) | 8 (13)
Anxiety (Psychiatric disorders) | 3 (3) | 6 (22)
ALT, SGPT (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Rigors/chills (General disorders) | 1 (1) | 5 (5)
Constipation (Gastrointestinal disorders) | 7 (17) | 11 (27)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (8)
Alkaline phosphatase (Metabolism and nutrition disorders) | 2 (5) | 0 (0)
Dehydration (Gastrointestinal disorders) | 1 (2) | 3 (5)
Depression (Psychiatric disorders) | 1 (1) | 2 (2)
Sweating (General disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 10 (32)
Dizziness (Nervous system disorders) | 4 (5) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 5 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 3 (6)
Edema - limb (Blood and lymphatic system disorders) | 1 (1) | 2 (3)
Erythema (Gastrointestinal disorders) | 3 (4) | 2 (3)
Fatigue (General disorders) | 7 (25) | 13 (67)
Fever (General disorders) | 2 (2) | 4 (4)
Hemoglobin (Blood and lymphatic system disorders) | 8 (29) | 14 (85)
Hot flashes (Endocrine disorders) | 1 (1) | 0 (0)
Bilirubin (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (9) | 4 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Infection NOS (Infections and infestations) | 1 (1) | 0 (0)
Infection - pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Infection - skin (Infections and infestations) | 1 (1) | 0 (0)
Infection - thrush (Infections and infestations) | 1 (1) | 2 (2)
Infection - upper respiratory (Infections and infestations) | 1 (1) | 0 (0)
Hypersensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Insomnia (General disorders) | 1 (1) | 5 (10)
Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Leukocytes (Blood and lymphatic system disorders) | 7 (24) | 15 (80)
Lymphopenia (Blood and lymphatic system disorders) | 2 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (18) | 14 (40)
Neuropathy (Nervous system disorders) | 2 (5) | 4 (18)
Neutrophils (ANC) (Blood and lymphatic system disorders) | 9 (25) | 16 (66)
Pain NOS (General disorders) | 3 (3) | 8 (23)
Pain - abdomen (General disorders) | 4 (6) | 9 (15)
Pain - back (General disorders) | 4 (8) | 4 (11)
Pain - bone (General disorders) | 2 (7) | 5 (65)
Pain - breast (General disorders) | 1 (1) | 0 (0)
Pain - chest (General disorders) | 2 (7) | 2 (3)
Pain - esophagus (General disorders) | 1 (1) | 2 (2)
Pain - joint (General disorders) | 4 (5) | 9 (34)
Pain - muscle (General disorders) | 2 (2) | 4 (8)
Pain - gums (General disorders) | 2 (2) | 0 (0)
Pain - stomach (General disorders) | 1 (1) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 1 (1) | 5 (28)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (14) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 1 (3) | 2 (5)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Weakness (General disorders) | 1 (1) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Hemorrhage NOS (Vascular disorders) | 1 (2) | 0 (0)
Pain - injection site (General disorders) | 1 (1) | 0 (0)
AST, SGPT (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Edema NOS (Blood and lymphatic system disorders) | 0 (0) | 3 (4)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (4)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (7)
Mucositis (Gastrointestinal disorders) | 0 (0) | 4 (7)
Pain - headache (General disorders) | 0 (0) | 8 (13)
Pain - limb (General disorders) | 0 (0) | 4 (4)
Pain - middle ear (General disorders) | 0 (0) | 2 (2)
Pain - mouth (General disorders) | 0 (0) | 2 (2)
Taste alteration (Gastrointestinal disorders) | 0 (0) | 2 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 9 (16)
Weight loss (General disorders) | 0 (0) | 2 (6)
Nasal reactions (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.